CLINICAL TRIAL: NCT03034356
Title: Reducing Hippocampal Hyperactivity and Improving Cognition in Schizophrenia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: MHBB-006-16S; I01CX001414 (NIH)
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Results first posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Levetiracetam, Then Placebo (Experimental): 4 weeks of levetiracetam administration (125 mg pill, bid), followed by a 4-week washout, then 4 weeks of placebo pill administration (bid).
  Interventions: Drug: Levetiracetam; Drug: Placebo
- Placebo, Then Levetiracetam (Experimental): 4 weeks of placebo administration (bid), followed by a 4-week washout, then 4 weeks of levetiracetam administration (125 mg pill, bid).
  Interventions: Drug: Levetiracetam; Drug: Placebo

INTERVENTIONS:
Drug: Levetiracetam — Anticonvulsant drug
  Other Names: Keppra
Drug: Placebo — Placebo

SUMMARY:
This study plans to learn more about the effects of levetiracetam (LEV) on brain activity and cognition in schizophrenia and schizoaffective disorder. Levetiracetam is an anti-seizure drug, also called an anticonvulsant.

DETAILED DESCRIPTION:
Cognitive symptoms are not currently well-managed in Veterans with schizophrenia, leading to substantially diminished quality of life. Improved treatment strategies clearly are needed. Recent studies suggest taht an overactive hippocampus is associated with cognitive deficits in the illness. Based on findings that the anti-epileptic drug levetiracetam (LEV) reduces hippocampal activity and improves cognition in other clinical populations while being safe and well-tolerated, this study will examine the effects of the drug on hippocampal activity and cognition in Veterans with schizophrenia. In this crossover design, participants will take LEV for 4 weeks and placebo pills for 4 weeks, but will not know the order in which they are taking them.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder
* Good general health
* Normal vital signs (blood pressure, pulse, respiration)

Exclusion Criteria:

* Substance abuse
* Significant neurological disorders
* Significant head trauma/injury
* Pregnancy
* MRI-specific exclusion criteria, e.g.,:

  * claustrophobia
  * weight>400 lbs
  * metal in the body

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason R. Tregellas, PhD, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be created and shared.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 67 patients were screened for eligibility between October 2018 and September 2023.
Pre-assignment Details: 41 out of 67 participants were randomized. Of those not randomized, 23 did not meet inclusion criteria and 3 declined to participate.
Period: Baseline
Arm/Group | Levetiracetam, Then Placebo | Placebo, Then Levetiracetam
Started | 20 | 21
Completed | 16 | 16
Not Completed | 4 | 5
Not completed — Lost to Follow-up | 2 | 4
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Physician Decision | 0 | 1
Period: Post-Intervention 1 (4 Weeks)
Arm/Group | Levetiracetam, Then Placebo | Placebo, Then Levetiracetam
Started | 16 | 16
Completed | 13 | 14
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Physician Decision | 1 | 0
Period: Post-Washout (4 Weeks)
Arm/Group | Levetiracetam, Then Placebo | Placebo, Then Levetiracetam
Started | 13 | 14
Completed | 11 | 14
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: Post-Intervention 2 (4 Weeks)
Arm/Group | Levetiracetam, Then Placebo | Placebo, Then Levetiracetam
Started | 11 | 14
Completed | 11 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levetiracetam, Then Placebo | Placebo, Then Levetiracetam | Total
Number analyzed (Participants) | 11 | 14 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.82 (16.65) | 48.00 (14.03) | 47.04 (14.95)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 8 | 10 | 18
  Other | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 8 | 10 | 18
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 4 | 6
  White | 9 | 7 | 16
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 11 | 14 | 25

OUTCOME MEASURES:

1. Primary Outcome: Neurocognitive Function
Description: Cognitive function as measured by the Repeatable Battery for the Assessment of Neurological Status (RBANS; total score). Scores are scaled with a mean of 100 and standard deviation of 15 (higher scores indicating better outcome).
Time Frame: 4 weeks
Population: All participants who received at least one dose of each intervention and completed all study visits were included.
Measure: Mean (Standard Deviation); unit: Total score
Groups:
- Levetiracetam: Participants who received levetiracetam administration (125 mg pill, bid) for either the first or last 4 weeks of the study.
- Placebo: Participants who received placebo administration (125 mg pill, bid) for either the first or last 4 weeks of the study.
Arm/Group | Levetiracetam | Placebo
Number analyzed (Participants) | 25 | 25
Total score
  RBANS at Baseline | 73.68 (14.69) | 74.04 (12.02)
  Change from Baseline at 4 weeks | 3.36 (7.29) | 3.96 (6.33)

2. Secondary Outcome: Resting-state Neuronal Response
Description: Neuronal response (measured via functional magnetic resonance imaging, fMRI) in the hippocampus during rest.
Time Frame: 4 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 4 weeks for each intervention
Description: All participants who received at least one dose of intervention.
Arm/Group | Levetiracetam | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/27
Other Adverse Events (participants affected / at risk) | 16/30 | 16/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Levetiracetam (N=30) | Placebo (N=27)
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Hallucinations (Psychiatric disorders) | 1 | 3
Headache (Nervous system disorders) | 3 | 2
Irritability (Psychiatric disorders) | 3 | 0
Paranoia (Psychiatric disorders) | 1 | 3
Sedation or Drowsiness (General disorders) | 6 | 3
Visual Disturbance (Eye disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT03034356/Prot_SAP_000.pdf